CLINICAL TRIAL: NCT05605548
Title: The Influence of Mitochondrial Derived Reactive Oxygen Species on Cardiovascular Health in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Mitochondrial Derived Reactive Oxygen Species on Cardiovascular Health in Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding was inconsistent and the Post-Doc left before the project ended
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20021976; 905812 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: MitoQ; vascular function; cardiovascular health; exercise intolerance; Mitochondria
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MitoQ (Experimental): Participants will take 1 pill each day for 6 weeks
  Interventions: Drug: MitoQ
- Placebo (Placebo Comparator): Participants will take 1 pill each day for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MitoQ — MitoQ is a mitochondrial targeted antioxidant that can be obtained over-the-counter.
  Arms: MitoQ
Other: Placebo — A look-alike inactive substance, a "sugar pill"
  Arms: Placebo

SUMMARY:
Cardiovascular health is a critical problem in patients with chronic obstructive pulmonary disease (COPD). Existing literature suggests oxidative stress from the mitochondria c driving some of the poor health outcomes in COPD. MitoQ is a mitochondrial-targeted antioxidant that has shown promise in improving cardiovascular outcomes in similar populations. Thus the purpose of this study is to test if MitoQ can improve cardiovascular health in COPD.

DETAILED DESCRIPTION:
In this study, a mitochondria-specific antioxidant will be compared to a placebo. Participants will be assigned randomly to receive either the antioxidant or the placebo for 6 weeks. A comprehensive assessment of cardiovascular health will be conducted before and after the administration of the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed of COPD
* Global Initiative for obstructive lung disease (GOLD) Stages II to IV

Exclusion Criteria:

* Forced Expiratory Volume in 1 second/ Functional Vital Capacity (FEV1/FVC) >0.7
* Heart Disease
* Diabetes
* Vasoactive medications
* Uncontrolled high blood pressure
* Fluid in lungs
* Sleep apnea
* Raynaud's Phenomenon
* Gangrene of the digits
* History of coagulation
* Pregnant women
* Children

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in vascular function | Baseline and 6 weeks
  Flow-mediated dilation will be used to measure vasodilation in the brachial artery
Change in Skeletal Muscle Oxygenation | Baseline and 6 weeks
  Near-infrared spectroscopy will be used to measure leg muscle oxygenation
Change in oxidative stress | Baseline and 6 weeks
  Blood draws will be taken to measure oxidative stress markers in the blood through electron paramagnetic resonance

SECONDARY OUTCOMES:
Change in arterial stiffness | Baseline and 6 weeks
  Pulse wave velocity will be used to measure arterial stiffness.
Change in microvascular function | Baseline and 6 weeks
  Microvascular function will be assessed using laser dopler imaging

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodriguez-Miguelez, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No